CLINICAL TRIAL: NCT02968849
Title: A Pivotal Phase 2b/3 Multisite, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of ALVAC-HIV (vCP2438) and Bivalent Subtype C gp120/MF59 in Preventing HIV-1 Infection in Adults in South Africa
Brief Title: Pivotal Phase 2b/3 ALVAC/Bivalent gp120/MF59 HIV Vaccine Prevention Safety and Efficacy Study in South Africa
Acronym: HVTN702
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanofi (Industry); GlaxoSmithKline (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 702
Record Dates: First submitted 2016-11-01; First posted 2016-11-21 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- ALVAC-HIV + subtype C gp120/MF59 (Active Comparator): 2700 participants will receive an IM injection of ALVAC-HIV (vCP2438) at months 0 and 1, and an IM injection of ALVAC-HIV (vCP2438) + Bivalent Subtype C gp120/MF59 at months 3, 6, and 12.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent Subtype C gp120/MF59
- Placebo (Placebo Comparator): 2700 participants will receive Sodium Chloride for injection, 0.9% at months 0, 1, 3, 6, and 12.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALVAC-HIV (vCP2438) — Expresses the gene products ZM96 gp120 (clade C strain) linked to the sequences encoding the HIV-1 transmembrane anchor (TM) sequence of gp41 (28 amino acids clade B LAI strain) and gag and pro (clade B LAI strain). It is formulated as a lyophilized vaccine for injection at a dose > 10^6 cell culture infectious dose 50% (CCIDv50) and < 1 × 10^8 CCIDv50 (nominal dose of 10^7 CCIDv50) and is reconstituted with 1 mL of sterile sodium chloride solution (NaCl 0.4%) delivered IM
  Arms: ALVAC-HIV + subtype C gp120/MF59
Biological: Bivalent Subtype C gp120/MF59 — Subtype C TV1.C gp120 Env and 1086.C gp120 Env proteins, each at a dose of 100 mcg, mixed with MF59 adjuvant (an oil-in-water emulsion) and delivered IM
  Arms: ALVAC-HIV + subtype C gp120/MF59
Biological: Placebo — Sodium Chloride for injection, 0.9% delivered IM
  Arms: Placebo

SUMMARY:
This study will evaluate the preventive vaccine efficacy, safety, and tolerability of ALVAC-HIV (vCP2438) + Bivalent Subtype C gp120/MF59 in HIV-seronegative South African adults over 24 months and potentially up to 36 months from enrollment.

DETAILED DESCRIPTION:
This study will evaluate the preventive vaccine efficacy, safety, and tolerability of the ALVAC-HIV vaccine + Bivalent Subtype C gp120 protein adjuvanted with MF59 in HIV-seronegative South African adults over 24 months from enrollment.

Participants will be randomized to receive ALVAC-HIV (vCP2438), or placebo, by intramuscular injection at weeks 0 and 4; they will receive ALVAC-HIV (vCP2438) + Bivalent Subtype C gp120/MF59, or placebo, by IM injection at weeks 12, 24, and 52.

In addition to the vaccination visits, participants will attend study visits at weeks 26, 39, 54, 65, 78, 91, 104, 117, 130, 142, and 156. All study visits, including vaccination visits, will include HIV risk reduction counseling, a physical exam, and an interview/questionnaire. and pregnancy testing for participants capable of becoming pregnant. Select study visits will include a medical history review, physical exam, blood collection, urine collection, HIV testing, and pregnancy testing for participants capable of becoming pregnant.

As of February 3, 2020, vaccinations for this study were suspended. Participants have been asked to continue attending follow-up visits for 12 months after the last vaccination they received. Participants who become HIV infected will be followed for 6 months after diagnosis.

ELIGIBILITY:
Inclusion Criteria

* Age of 18 to 35 years
* Sexually active, defined as having had sexual intercourse at least twice in the past 30 days prior to screening, and is considered by the site staff to be at risk for HIV infection.
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study prior to first vaccination with verbal demonstration of understanding of all questions.
* Agrees not to enroll in another study of an investigational research agent until the participant is unblinded or their study participation ends, whichever occurs last
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and willing to receive HIV risk reduction counseling.
* Alanine aminotransferase (ALT) < 2.5 times the institutional upper limit of normal
* Negative HIV-1 and -2 blood test within 30 days prior to enrollment: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (Appendix B and Appendix C) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through 3 months after the last vaccination. Effective contraception is defined as using 2 methods of birth control. These include 1 of the following methods:

    * Condoms (male or female)
    * Diaphragm or cervical cap

PLUS 1 of the following methods:

* Intrauterine device (IUD),
* Hormonal contraception (in accordance with applicable national contraception guidelines), or
* Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy), or
* Any other contraceptive method approved by the protocol safety review team;

  * Or not be of reproductive potential, such as having been diagnosed with premature menopause (with no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.

    * Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until 3 months after the last vaccination

Exclusion Criteria

* Blood products received within 90 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the study
* Pregnant or breastfeeding
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 702 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure. For volunteers who have received control/placebo in an experimental vaccine trial, the protocol safety review team will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the protocol safety review team on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Immunosuppressive medications received within 168 days before first vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components such as eggs, egg products, or neomycin including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a non-anaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Immunodeficiency
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Active tuberculosis (TB) disease
* Uncontrolled hypertension: systolic blood pressure (SBP) ≥ 160 mm Hg or diastolic blood pressure (DBP) ≥ 100 mm Hg
* Bleeding disorder (diagnosed by a doctor) contraindicating IM injection and/or blood draws, based on investigator's judgment
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5404 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, MD, Study Chair — Perinatal HIV Research Unit (PHRU), Chris Hani Baragwanath Hospital
Locations (14):
- South Africa (14):
  - Walter Sisulu University HIV Vaccine Research Unit CRS, Mthatha, Eastern Cape
  - Kliptown Soweto CRS, Johannesburg, Gauteng
  - Aurum Tembisa CRS, Johannesburg, Gauteng
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - MeCRU CRS, Pretoria, Gauteng
  - Setshaba Research Centre CRS, Soshanguve, Gauteng
  - eThekwini CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Isipingo, KwaZulu-Natal
  - Qhakaza Mbokodo Research Clinic CRS, Ladysmith, KwaZulu-Natal
  - Verulam CRS, Verulam, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Rustenburg CRS, Rustenburg, North West
  - Emavundleni CRS, Cape Town, Western Cape
  - Khayelitsha CRS, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray GE, Bekker LG, Laher F, Malahleha M, Allen M, Moodie Z, Grunenberg N, Huang Y, Grove D, Prigmore B, Kee JJ, Benkeser D, Hural J, Innes C, Lazarus E, Meintjes G, Naicker N, Kalonji D, Nchabeleng M, Sebe M, Singh N, Kotze P, Kassim S, Dubula T, Naicker V, Brumskine W, Ncayiya CN, Ward AM, Garrett N, Kistnasami G, Gaffoor Z, Selepe P, Makhoba PB, Mathebula MP, Mda P, Adonis T, Mapetla KS, Modibedi B, Philip T, Kobane G, Bentley C, Ramirez S, Takuva S, Jones M, Sikhosana M, Atujuna M, Andrasik M, Hejazi NS, Puren A, Wiesner L, Phogat S, Diaz Granados C, Koutsoukos M, Van Der Meeren O, Barnett SW, Kanesa-Thasan N, Kublin JG, McElrath MJ, Gilbert PB, Janes H, Corey L; HVTN 702 Study Team. Vaccine Efficacy of ALVAC-HIV and Bivalent Subtype C gp120-MF59 in Adults. N Engl J Med. 2021 Mar 25;384(12):1089-1100. doi: 10.1056/NEJMoa2031499. PMID 33761206
- [Background] Moodie Z, Dintwe O, Sawant S, Grove D, Huang Y, Janes H, Heptinstall J, Omar FL, Cohen K, De Rosa SC, Zhang L, Yates NL, Sarzotti-Kelsoe M, Seaton KE, Laher F, Bekker LG, Malahleha M, Innes C, Kassim S, Naicker N, Govender V, Sebe M, Singh N, Kotze P, Lazarus E, Nchabeleng M, Ward AM, Brumskine W, Dubula T, Randhawa AK, Grunenberg N, Hural J, Kee JJ, Benkeser D, Jin Y, Carpp LN, Allen M, D'Souza P, Tartaglia J, DiazGranados CA, Koutsoukos M, Gilbert PB, Kublin JG, Corey L, Andersen-Nissen E, Gray GE, Tomaras GD, McElrath MJ. Analysis of the HIV Vaccine Trials Network 702 Phase 2b-3 HIV-1 Vaccine Trial in South Africa Assessing RV144 Antibody and T-Cell Correlates of HIV-1 Acquisition Risk. J Infect Dis. 2022 Aug 24;226(2):246-257. doi: 10.1093/infdis/jiac260. PMID 35758878
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Chihana R, Jin Kee J, Moodie Z, Huang Y, Janes H, Dadabhai S, Roxby AC, Allen M, Kassim S, Naicker V, Innes C, Naicker N, Dubula T, Grunenberg N, Malahleha M, Kublin JG, Bekker LG, Gray G, Kumwenda J, Laher F. Factors associated with reactogenicity to an investigational HIV vaccine regimen in HIV vaccine trials network 702. Vaccine. 2024 Aug 13;42(20):125991. doi: 10.1016/j.vaccine.2024.05.039. Epub 2024 May 21. PMID 38772835
- [Derived] Laher F, Malahleha M, Ramirez S, Brumskine W, Otwombe K, Moodie Z, Allen M. Data quality in an HIV vaccine efficacy clinical trial in South Africa: through natural disasters and with discipline. BMC Med Res Methodol. 2023 Jun 24;23(1):147. doi: 10.1186/s12874-023-01967-9. PMID 37355583
- [Derived] Hanass-Hancock J, Carpenter B, Reddy T, Nzuza A, Gaffoor Z, Goga A, Andrasik M. Participants' characteristics and motivations to screen for HIV vaccine and monoclonal antibody trials in KwaZulu-Natal, South Africa. Trials. 2021 Dec 11;22(1):897. doi: 10.1186/s13063-021-05792-7. PMID 34895272

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: ALVAC-HIV at months 0, 1, 3, 6, 12, 18, and bivalent subtype C gp120/MF9 at months 3, 6, 12, 18
- Placebo: Placebo for ALVAC-HIV at months 0, 1, 3, 6, 12, 18, and placebo for bivalent subtype C gp120/MF9 at months 3, 6, 12, 18
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 2704 | 2700
Modified Intent-to-Treat (MITT) Cohort | 2695 | 2689
MITT Infected Cohort | 151 | 143
Week 26 At-Risk Cohort | 2430 | 2393
Immunogenicity Cohort | 120 | 10
Completed | 2557 | 2557
Not Completed | 147 | 143
Not completed — Death | 8 | 10
Not completed — Lost to Follow-up | 31 | 29
Not completed — Withdrawal by Subject | 73 | 64
Not completed — Participant Unable to Adhere to Visit Schedule | 13 | 21
Not completed — Physician Decision | 6 | 9
Not completed — Other | 16 | 10

BASELINE CHARACTERISTICS:
Population: Safety Cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 2704 | 2700 | 5404
Age, Continuous [Median (Full Range); unit: Years]
  Female | 24 [18 to 35] | 23 [18 to 35] | 24 [18 to 35]
  Male | 26 [18 to 35] | 26 [18 to 35] | 26 [18 to 35]
Age, Customized [Count of Participants; unit: Participants] — Population: Age categories are summarized separately within females and males.
  Participants
    Female: number analyzed (Participants) | 1893 | 1893 | 3786
    Female: 18 - 20 years | 349 | 392 | 741
    Female: 21 - 25 years | 917 | 877 | 1794
    Female: 26 - 30 years | 465 | 461 | 926
    Female: 31 - 35 years | 162 | 163 | 325
    Male: number analyzed (Participants) | 811 | 807 | 1618
    Male: 18 - 20 years | 114 | 98 | 212
    Male: 21 - 25 years | 271 | 276 | 547
    Male: 26 - 30 years | 244 | 254 | 498
    Male: 31 - 35 years | 182 | 179 | 361
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1893 | 1893 | 3786
  Male | 811 | 807 | 1618
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2704 | 2700 | 5404
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2672 | 2676 | 5348
  Colored/Mixed | 23 | 17 | 40
  White | 3 | 3 | 6
  Indian | 1 | 1 | 2
  Asian | 0 | 1 | 1
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  South Africa | 2704 | 2700 | 5404

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment (Concurrent With First Vaccination) Through 24 Months After Enrollment
Description: Vaccine efficacy was calculated as 1 minus the hazard ratio for HIV-1 infection, which was estimated using a sex-stratified Cox proportional-hazards (Cox PH) model and tested using a sex-stratified log-rank test. Vaccine efficacy was also measured using a ratio of cumulative incidences (CIR) of HIV-1 infection in the vaccine group as compared with the placebo group, which was calculated using Nelson-Aalen cumulative hazard estimates and tested using a Wald test.
Time Frame: Measured through 24 months after first vaccination
Population: MITT cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2695 | 2689
events per 100 person-years
  Cox PH method | 0.034 | 0.033
  CIR method | 0.034 | 0.033
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.84, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.81 to 1.30] — The hazard ratio was estimated using a sex-stratified Cox proportional hazards model. The vaccine group (ALVAC-HIV + subtype C gp120/MF59) represents the numerator and the placebo group represents the denominator
Statistical Analysis 2: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.83, Wald; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.81 to 1.31] — The hazard ratio was estimated using Nelson-Aalen cumulative hazard estimates. The vaccine group (ALVAC-HIV + subtype C gp120/MF59) represents the numerator and the placebo group represents the denominator

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 full days following each vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Pain: None | 2161 | 2539
  Pain: Mild | 480 | 149
  Pain: Moderate | 62 | 12
  Pain: Severe | 1 | 0
  Pain: Potentially Life-threatening | 0 | 0
  Tenderness: None | 2368 | 2600
  Tenderness: Mild | 297 | 91
  Tenderness: Moderate | 38 | 9
  Tenderness: Severe | 1 | 0
  Tenderness: Potentially Life-threatening | 0 | 0
  Pain and/or Tenderness: None | 2082 | 2493
  Pain and/or Tenderness: Mild | 552 | 194
  Pain and/or Tenderness: Moderate | 69 | 13
  Pain and/or Tenderness: Severe | 1 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0

3. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 2
Time Frame: Measured through 3 full days following each vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Erythema/Redness: None / Not Gradable | 2494 | 2683
  Erythema/Redness: Gr 1: 2.5 - <5cm / 6.25 - <25cm^2 | 108 | 14
  Erythema/Redness: Gr 2: 5 - <10cm / 25 - <100cm^2 | 74 | 3
  Erythema/Redness: Gr 3: >=10cm / >=100cm^2 / Complications | 28 | 0
  Erythema/Redness: Gr 4: Complications | 0 | 0
  Induration/Swelling: None / Not Gradable | 2380 | 2675
  Induration/Swelling: Gr 1: 2.5 - <5cm / 6.25 - <25cm^2 | 159 | 16
  Induration/Swelling: Gr 2: 5 - <10cm / 25 - <100cm^2 | 133 | 7
  Induration/Swelling: Gr 3: >=10cm / >=100cm^2 / Complications | 32 | 2
  Induration/Swelling: Gr 4: Complications | 0 | 0
  Erythema and/or Induration: None / Not Gradable | 2314 | 2662
  Erythema and/or Induration: Gr 1: 2.5 - <5cm / 6.25 - <25cm^2 | 196 | 26
  Erythema and/or Induration: Gr 2: 5 - <10cm / 25 - <100cm^2 | 156 | 10
  Erythema and/or Induration: Gr 3: >=10cm / >=100cm^2 / Complications | 38 | 2
  Erythema and/or Induration: Gr 4: Complications | 0 | 0

4. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 2
Time Frame: Measured through 3 full days following each vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Arthralgia: None | 2622 | 2649
  Arthralgia: Mild | 75 | 40
  Arthralgia: Moderate | 7 | 11
  Arthralgia: Severe | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0
  Arthralgia: Missing | 0 | 0
  Chills: None | 2614 | 2641
  Chills: Mild | 87 | 51
  Chills: Moderate | 3 | 8
  Chills: Severe | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0
  Chills: Missing | 0 | 0
  Headache: None | 2267 | 2276
  Headache: Mild | 317 | 311
  Headache: Moderate | 117 | 112
  Headache: Severe | 3 | 1
  Headache: Potentially Life-threatening | 0 | 0
  Headache: Missing | 0 | 0
  Malaise and/or fatigue: None | 2461 | 2497
  Malaise and/or fatigue: Mild | 221 | 177
  Malaise and/or fatigue: Moderate | 21 | 24
  Malaise and/or fatigue: Severe | 1 | 2
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Malaise and/or fatigue: Missing | 0 | 0
  Myalgia: None | 2604 | 2644
  Myalgia: Mild | 85 | 48
  Myalgia: Moderate | 15 | 8
  Myalgia: Severe | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0
  Myalgia: Missing | 0 | 0
  Nausea: None | 2585 | 2583
  Nausea: Mild | 104 | 107
  Nausea: Moderate | 15 | 10
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Nausea: Missing | 0 | 0
  Vomiting: None | 2625 | 2629
  Vomiting: Mild | 64 | 64
  Vomiting: Moderate | 15 | 7
  Vomiting: Severe | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0
  Vomiting: Missing | 0 | 0
  Max. Systemic Symptoms (excl. Temp.): None | 2004 | 2095
  Max. Systemic Symptoms (excl. Temp.): Mild | 545 | 459
  Max. Systemic Symptoms (excl. Temp.): Moderate | 151 | 143
  Max. Systemic Symptoms (excl. Temp.): Severe | 4 | 3
  Max. Systemic Symptoms (excl. Temp.): Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms (excl. Temp.): Missing | 0 | 0
  Temperature: None | 2409 | 2406
  Temperature: Mild | 168 | 176
  Temperature: Moderate | 98 | 84
  Temperature: Severe | 19 | 15
  Temperature: Potentially Life-threatening | 1 | 5
  Temperature: Missing | 9 | 14

5. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Relationship to Study Product
Description: For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through 30 days after each vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Related | 38 | 12
  Not Related | 1689 | 1722
  No AE Reported | 977 | 966

6. Primary Outcome: Number of Participants Reporting Adverse Events (AEs), by Severity Grade
Description: For participants reporting multiple AEs over the time frame, the maximum severity grade is counted.
Time Frame: Measured through 30 days after each vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Mild | 161 | 137
  Moderate | 1443 | 1472
  Severe | 98 | 103
  Potentially life-threatening | 17 | 12
  Death | 8 | 10
  No AE Reported | 977 | 966

7. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: Measured as outlined in Version 2.0 (January 2010) of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual).
Time Frame: Measured through 12 months after last vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Yes | 103 | 95
  No | 1624 | 1639
  No AE Reported | 977 | 966

8. Primary Outcome: Number of Participants Reporting Adverse Events of Special Interest (AESIs)
Description: Adverse events of special interest (AESI) were described in Appendix J of the protocol. AESI for this protocol include but are not limited to potential immune-mediated diseases.
Time Frame: Measured through 12 months after last vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Yes | 4 | 2
  No | 1693 | 1700
  No AE Reported | 1007 | 998

9. Primary Outcome: Number of Participants Reporting New Chronic Medical Conditions
Description: A new chronic medical condition is defined as a new onset or exacerbation of medical condition requiring 2 or more visits to a medical provider during a period of at least 30 days.
Time Frame: Measured through 12 months after last vaccination
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Yes | 54 | 54
  No | 1673 | 1680
  No AE Reported | 977 | 966

10. Primary Outcome: Number of Participants With Early Study Termination Associated With an AE or Reactogenicity
Description: From the termination form, early study termination associated with an AE or reactogenicity reasons are tabulated by treatment group.
Time Frame: Measured through study completion (through 6 months after confirmation of HIV-1 diagnosis for participants who acquired HIV and through 12 months after last vaccination for the rest)
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Termination associated with adverse event or reactogenicity | 9 | 14
  Other reason | 140 | 129
  No discontinuation | 2555 | 2557

11. Primary Outcome: Number of Participants With Study Product Discontinuation Associated With an AE or Reactogenicity
Description: From the study product discontinuation form, study product discontinuation reasons are tabulated by treatment group.
Time Frame: as for outcome 10
Population: Safety cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2704 | 2700
Participants
  Clinical event other than reactogenicity, HIV, infection or death | 8 | 6
  Reactogenicity symptom | 4 | 1
  Other reason | 539 | 598
  No discontinuation | 2153 | 2095

12. Primary Outcome: Incidence Rate of HIV-1 Infections Diagnosed Following Enrollment and Throughout All Participant Follow-Up
Description: Per the 23 January 2020 DSMB finding that monitoring boundaries for non-efficacy have been met, Primary outcome 1 has been superseded by this primary outcome. Vaccine efficacy was calculated as 1 minus the hazard ratio for HIV-1 infection, which was estimated using a sex-stratified Cox proportional-hazards (Cox PH) model and tested using a sex-stratified log-rank test. Vaccine efficacy was also measured using a ratio of cumulative incidences (CIR) of HIV-1 infection in the vaccine group as compared with the placebo group, which was calculated using Nelson-Aalen cumulative hazard estimates and tested using a Wald test.
Time Frame: Measured through 36 months after first vaccination
Population: MITT cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2695 | 2689
events per 100 person-years
  Cox PH method | 0.032 | 0.03
  CIR method | 0.038 | 0.03
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.66, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.85 to 1.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.98, Wald; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.81 to 1.23] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through 36 Months Post Enrollment
Description: This outcome measure is the same as Primary Outcome 12, which was added after pre-established criteria for vaccine non-efficacy had been met. Analysis was not repeated but the outcome is listed for completeness.
Time Frame: Measured through 36 months after first vaccination
Population: This outcome measure is the same as Primary Outcome 12, which was added after pre-established criteria for vaccine non-efficacy had been met. Analysis was not repeated but the outcome is listed for completeness.
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Month 6.5 Through 24 Months Post Enrollment
Description: as for outcome 1
Time Frame: Measured after Month 6.5 through 24 months after first vaccination
Population: Week 26 at-risk cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2430 | 2393
events per 100 person-years
  Cox PH method | 0.03 | 0.026
  CIR method | 0.03 | 0.026
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.39, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.84 to 1.58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.50, Wald; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.81 to 1.54] — [estimate comment as in outcome 1, analysis 2]

15. Secondary Outcome: Number of Participants With Occurrence of CD4+ and CD8+ T-Cells Expressing IFN-g and/or IL-2 in Response to HIV Proteins Included in the Vaccine at Month 6.5
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as negative control. Response magnitude is % cells expressing IFN-g and/or IL-2 after stimulation minus % cells expressing markers after no stimulation. Contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). One-sided Fisher's exact test is applied, testing if number of cells positive for the marker is equal in stimulated vs. unstimulated cells. Bonferroni-Holm adjustment is made over peptide pools. Response is positive if adjusted p-value le 0.00001. Data are excluded if blood draw date was outside visit window, participant was HIV-infected (post-infection samples), PBMC viability/T-cell count were low or negative control was high. Any Env is the maximum of ZM96 gp120, 1086 gp120, and TV1 gp120. Any HIV is the sum of Any Env and LAI Gag. Negative magnitudes are censored at 0 before calculating sum; if the sum is lt 0.01, it is set to 0.01%.
Time Frame: Measured at Month 6.5
Population: Immunogenicity cohort. "Overall Number of Participants Analyzed" represents participants in the immunogenicity cohort who have samples collected at Month 6.5 and who were HIV-uninfected. "Number Analyzed" represents those participants with available data after filtering for assay-specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 119 | 10
Participants
  CD4+ : 1086 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : 1086 gp120 | 65 | 0
  CD4+ : ANY ENV: number analyzed (Participants) | 117 | 10
  CD4+ : ANY ENV | 88 | 0
  CD4+ : ANY HIV: number analyzed (Participants) | 117 | 10
  CD4+ : ANY HIV | 89 | 0
  CD4+ : LAI Gag: number analyzed (Participants) | 117 | 10
  CD4+ : LAI Gag | 4 | 0
  CD4+ : TV1 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : TV1 gp120 | 86 | 0
  CD4+ : ZM96 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : ZM96 gp120 | 78 | 0
  CD8+ : 1086 gp120: number analyzed (Participants) | 118 | 10
  CD8+ : 1086 gp120 | 2 | 0
  CD8+ : ANY ENV: number analyzed (Participants) | 118 | 10
  CD8+ : ANY ENV | 13 | 0
  CD8+ : ANY HIV: number analyzed (Participants) | 118 | 10
  CD8+ : ANY HIV | 15 | 0
  CD8+ : LAI Gag: number analyzed (Participants) | 117 | 10
  CD8+ : LAI Gag | 4 | 0
  CD8+ : TV1 gp120: number analyzed (Participants) | 118 | 10
  CD8+ : TV1 gp120 | 4 | 0
  CD8+ : ZM96 gp120: number analyzed (Participants) | 117 | 10
  CD8+ : ZM96 gp120 | 11 | 0

16. Secondary Outcome: Number of Participants With Occurrence of CD4+ and CD8+ T-Cells Expressing IFN-g and/or IL-2 and/or CD40L in Response to HIV Proteins Included in the Vaccine at Month 6.5
Description: as for outcome 15
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 119 | 10
Participants
  CD4+ : 1086 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : 1086 gp120 | 86 | 0
  CD4+ : ANY ENV: number analyzed (Participants) | 117 | 10
  CD4+ : ANY ENV | 103 | 0
  CD4+ : ANY HIV: number analyzed (Participants) | 117 | 10
  CD4+ : ANY HIV | 103 | 0
  CD4+ : LAI Gag: number analyzed (Participants) | 117 | 10
  CD4+ : LAI Gag | 7 | 0
  CD4+ : TV1 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : TV1 gp120 | 99 | 0
  CD4+ : ZM96 gp120: number analyzed (Participants) | 117 | 10
  CD4+ : ZM96 gp120 | 88 | 0
  CD8+ : 1086 gp120: number analyzed (Participants) | 118 | 10
  CD8+ : 1086 gp120 | 5 | 0
  CD8+ : ANY ENV: number analyzed (Participants) | 118 | 10
  CD8+ : ANY ENV | 16 | 0
  CD8+ : ANY HIV: number analyzed (Participants) | 118 | 10
  CD8+ : ANY HIV | 17 | 0
  CD8+ : LAI Gag: number analyzed (Participants) | 117 | 10
  CD8+ : LAI Gag | 3 | 0
  CD8+ : TV1 gp120: number analyzed (Participants) | 118 | 10
  CD8+ : TV1 gp120 | 6 | 0
  CD8+ : ZM96 gp120: number analyzed (Participants) | 117 | 10
  CD8+ : ZM96 gp120 | 11 | 0

17. Secondary Outcome: Level of CD4+ and CD8+ T-Cells Expressing IFN-g and/or IL-2 in Response to HIV Proteins Included in the Vaccine at Month 6.5
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as negative control. Response magnitude is % cells expressing IFN-g and/or IL-2 after stimulation minus % cells expressing markers after no stimulation. Data are excluded if blood draw date was outside visit window, participant was HIV-infected (post-infection samples), PBMC viability/T-cell count were low or negative control was high. Any Env is the maximum of ZM96 gp120, 1086 gp120, and TV1 gp120. Any HIV is the sum of Any Env and LAI Gag. Negative magnitudes are censored at 0 before calculating sum; if the sum is lt 0.01, it is set to 0.01%. Summary was calculated among positive responders only.
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: % T-Cells
Arm/Group | Vaccine
Number analyzed (Participants) | 119
% T-Cells
  CD4+ : 1086 gp120: number analyzed (Participants) | 65
  CD4+ : 1086 gp120 | 0.1 [0.1 to 0.2]
  CD4+ : ANY ENV: number analyzed (Participants) | 88
  CD4+ : ANY ENV | 0.1 [0.1 to 0.2]
  CD4+ : ANY HIV: number analyzed (Participants) | 89
  CD4+ : ANY HIV | 0.2 [0.1 to 0.2]
  CD4+ : LAI Gag: number analyzed (Participants) | 4
  CD4+ : LAI Gag | 0.1 [0 to 0.1]
  CD4+ : TV1 gp120: number analyzed (Participants) | 86
  CD4+ : TV1 gp120 | 0.1 [0.1 to 0.2]
  CD4+ : ZM96 gp120: number analyzed (Participants) | 78
  CD4+ : ZM96 gp120 | 0.1 [0.1 to 0.2]
  CD8+ : 1086 gp120: number analyzed (Participants) | 2
  CD8+ : 1086 gp120 | 0.1 [0.1 to 0.1]
  CD8+ : ANY ENV: number analyzed (Participants) | 13
  CD8+ : ANY ENV | 0.1 [0.1 to 0.2]
  CD8+ : ANY HIV: number analyzed (Participants) | 15
  CD8+ : ANY HIV | 0.1 [0.1 to 0.2]
  CD8+ : LAI Gag: number analyzed (Participants) | 4
  CD8+ : LAI Gag | 0.1 [0.1 to 0.2]
  CD8+ : TV1 gp120: number analyzed (Participants) | 4
  CD8+ : TV1 gp120 | 0.1 [0.1 to 0.1]
  CD8+ : ZM96 gp120: number analyzed (Participants) | 11
  CD8+ : ZM96 gp120 | 0.1 [0.1 to 0.2]

18. Secondary Outcome: Level of CD4+ and CD8+ T-Cells Expressing IFN-g and/or IL-2 and/or CD40L in Response to HIV Proteins Included in the Vaccine at Month 6.5
Description: as for outcome 17
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: % T-Cells
Arm/Group | Vaccine
Number analyzed (Participants) | 119
% T-Cells
  CD4+ : 1086 gp120: number analyzed (Participants) | 86
  CD4+ : 1086 gp120 | 0.2 [0.1 to 0.3]
  CD4+ : ANY ENV: number analyzed (Participants) | 103
  CD4+ : ANY ENV | 0.2 [0.1 to 0.3]
  CD4+ : ANY HIV: number analyzed (Participants) | 103
  CD4+ : ANY HIV | 0.2 [0.2 to 0.4]
  CD4+ : LAI Gag: number analyzed (Participants) | 7
  CD4+ : LAI Gag | 0.1 [0.1 to 0.1]
  CD4+ : TV1 gp120: number analyzed (Participants) | 99
  CD4+ : TV1 gp120 | 0.2 [0.1 to 0.3]
  CD4+ : ZM96 gp120: number analyzed (Participants) | 88
  CD4+ : ZM96 gp120 | 0.2 [0.1 to 0.3]
  CD8+ : 1086 gp120: number analyzed (Participants) | 5
  CD8+ : 1086 gp120 | 0.1 [0.1 to 0.1]
  CD8+ : ANY ENV: number analyzed (Participants) | 16
  CD8+ : ANY ENV | 0.1 [0.1 to 0.2]
  CD8+ : ANY HIV: number analyzed (Participants) | 17
  CD8+ : ANY HIV | 0.2 [0.1 to 0.2]
  CD8+ : LAI Gag: number analyzed (Participants) | 3
  CD8+ : LAI Gag | 0.1 [0.1 to 0.3]
  CD8+ : TV1 gp120: number analyzed (Participants) | 6
  CD8+ : TV1 gp120 | 0.1 [0.1 to 0.1]
  CD8+ : ZM96 gp120: number analyzed (Participants) | 11
  CD8+ : ZM96 gp120 | 0.1 [0.1 to 0.2]

19. Secondary Outcome: Number of Participants With Occurrence of Vaccine-induced IgG Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution.The readout is background-subtracted mean fluorescent intensity(MFI),with background adjustment for an antigen-specific plate level control.For each sample,response magnitude is net MFI,defined as experimental antigen MFI minus reference antigen MFI. Net MFI lt 1 is set to 1,and net MFI > 22,000 is set to 22,000.Data are excluded if blood draw date was outside the allowable window,a participant was HIV-infected,reference antigen > 5,000 MFI or baseline net MFI > 6,500.Samples from post-enrollment visits have positive responses if they meet three criteria:(1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI),(2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI.
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 120 | 10
Participants
  HVTN 505 Env Breadth Panel : VRC A_avi: number analyzed (Participants) | 117 | 10
  HVTN 505 Env Breadth Panel : VRC A_avi | 117 | 0
  HVTN 505 Env Breadth Panel : VRC B gp140: number analyzed (Participants) | 117 | 10
  HVTN 505 Env Breadth Panel : VRC B gp140 | 116 | 0
  HVTN 505 Env Breadth Panel : VRC C_avi: number analyzed (Participants) | 117 | 10
  HVTN 505 Env Breadth Panel : VRC C_avi | 117 | 0
  RV144 CoR IgA Primary gp120 Score : 00MSA 4076 gp140: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : 00MSA 4076 gp140 | 117 | 0
  RV144 CoR IgA Primary gp120 Score : A244 gp 120 gDneg/293F/mon: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : A244 gp 120 gDneg/293F/mon | 117 | 0
  RV144 CoR IgA Primary gp120 Score : B.con.env03 140 CF: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : B.con.env03 140 CF | 117 | 0
  RV144 CoR IgA Primary gp120 Score : C.con.env03 140 CF_avi: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : C.con.env03 140 CF_avi | 117 | 0
  RV144 CoR IgA Primary gp120 Score : Con 6 gp120/B: number analyzed (Participants) | 114 | 9
  RV144 CoR IgA Primary gp120 Score : Con 6 gp120/B | 114 | 0
  RV144 CoR IgA Primary gp120 Score : Con S gp140 CFI: number analyzed (Participants) | 114 | 9
  RV144 CoR IgA Primary gp120 Score : Con S gp140 CFI | 114 | 0
  RV144 CoR IgA Primary gp120 Score : G.con.env03 140 CF: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : G.con.env03 140 CF | 117 | 0
  RV144 CoR IgA Primary gp120 Score : HV 13700 AE.con.env03 140 CF: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : HV 13700 AE.con.env03 140 CF | 117 | 0
  RV144 CoR IgA Primary gp120 Score : HV 14000 (DRCBL) gp140: number analyzed (Participants) | 117 | 10
  RV144 CoR IgA Primary gp120 Score : HV 14000 (DRCBL) gp140 | 117 | 0
  RV144 CoR IgG : 92TH023 gp120 gDneg 293F mon: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : 92TH023 gp120 gDneg 293F mon | 117 | 0
  RV144 CoR IgG : A1.con.env03 140 CF: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : A1.con.env03 140 CF | 117 | 0
  RV144 CoR IgG : AE.A244 V1V2 Tags/293F: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : AE.A244 V1V2 Tags/293F | 103 | 0
  RV144 CoR IgG : C.1086C_V1_V2 Tags: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : C.1086C_V1_V2 Tags | 86 | 0
  RV144 CoR IgG : gp70-92TH023 V1V2: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : gp70-92TH023 V1V2 | 112 | 0
  RV144 CoR IgG : gp70_B.CaseA_V1_V2: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG : gp70_B.CaseA_V1_V2 | 62 | 0
  RV144 CoR IgG3 : gp70_B.CaseA2 V1/V2/169K: number analyzed (Participants) | 117 | 10
  RV144 CoR IgG3 : gp70_B.CaseA2 V1/V2/169K | 63 | 0
  RV144 CoR IgA : Bio-1086C C1_HS: number analyzed (Participants) | 116 | 10
  RV144 CoR IgA : Bio-1086C C1_HS | 59 | 0
  RV144 CoR IgA : Bio-92TH023 C1_HS: number analyzed (Participants) | 116 | 10
  RV144 CoR IgA : Bio-92TH023 C1_HS | 96 | 0
  RV144 CoR IgA : Bio-96ZM651 C1_HS: number analyzed (Participants) | 116 | 10
  RV144 CoR IgA : Bio-96ZM651 C1_HS | 92 | 0
  RV144 CoR IgA : Bio-TV1 C1_HS: number analyzed (Participants) | 116 | 10
  RV144 CoR IgA : Bio-TV1 C1_HS | 42 | 0
  Vaccine Matched Env : 1086C_D7gp120.avi/293F: number analyzed (Participants) | 114 | 9
  Vaccine Matched Env : 1086C_D7gp120.avi/293F | 114 | 0
  Vaccine Matched Env : 96ZM651.D11gp120.avi: number analyzed (Participants) | 113 | 9
  Vaccine Matched Env : 96ZM651.D11gp120.avi | 113 | 0
  Vaccine Matched Env : TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 114 | 9
  Vaccine Matched Env : TV1c8_D11gp120.avi/293F | 114 | 0
  Vaccine Strain Matched V1V2 : gp70-96ZM651.02 V1v2: number analyzed (Participants) | 116 | 10
  Vaccine Strain Matched V1V2 : gp70-96ZM651.02 V1v2 | 61 | 0
  Vaccine Strain Matched V1V2 : gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 117 | 10
  Vaccine Strain Matched V1V2 : gp70-TV1.GSKvacV1V2/293F | 73 | 0
  Vaccine Strain Matched V1V2 : gp70_C.1086C V1/V2/293F: number analyzed (Participants) | 117 | 10
  Vaccine Strain Matched V1V2 : gp70_C.1086C V1/V2/293F | 103 | 0
  gp41: number analyzed (Participants) | 117 | 10
  gp41 | 1 | 0

20. Secondary Outcome: Number of Participants With Occurrence of Vaccine-induced IgG3 Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgG3 responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay,run at 1:40 dilution.The readout is background-subtracted mean fluorescent intensity(MFI), with background adjustment for an antigen-specific plate level control.For each sample, response magnitude is net MFI,defined as experimental antigen MFI minus reference antigen MFI.Net MFI lt 1 is set to 1, and net MFI > 22,000 is set to 22,000.Data are excluded if blood draw date was outside the allowable window,a participant was HIV-infected,reference antigen > 5,000 MFI or baseline net MFI > 6,500.Samples from post-enrollment visits have positive responses if they meet three criteria:(1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), (2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline M
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 120 | 10
Participants
  HVTN 505 Env Breadth Panel : A1.con.env03 140 CF | 74 | 0
  HVTN 505 Env Breadth Panel : B.con.env03 140 CF | 106 | 0
  HVTN 505 Env Breadth Panel : C.con.env03 140 CF_avi | 87 | 0
  HVTN 505 Env Breadth Panel : Con 6 gp120/B | 99 | 0
  HVTN 505 Env Breadth Panel : Con S gp140 CFI | 115 | 0
  HVTN 505 Env Breadth Panel : VRC A_avi | 72 | 0
  HVTN 505 Env Breadth Panel : VRC B gp140 | 42 | 0
  HVTN 505 Env Breadth Panel : VRC C_avi | 68 | 0
  RV144 CoR IgG3 : C.1086C_V1_V2 Tags | 32 | 0
  RV144 CoR IgG3 : gp70_B.CaseA2 V1/V2/169K | 9 | 0
  RV144 CoR IgG3 : gp70_B.CaseA_V1_V2 | 8 | 0
  V1V2 Subtype AW : AE.A244 V1V2 Tags/293F | 49 | 0
  Vaccine Matched Env : 1086C_D7gp120.avi/293F | 120 | 0
  Vaccine Matched Env : 96ZM651.D11gp120.avi | 110 | 0
  Vaccine Matched Env : TV1c8_D11gp120.avi/293F | 118 | 0
  Vaccine Strain Matched V1V2 : gp70-96ZM651.02 V1v2: number analyzed (Participants) | 118 | 10
  Vaccine Strain Matched V1V2 : gp70-96ZM651.02 V1v2 | 10 | 0
  Vaccine Strain Matched V1V2 : gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 118 | 10
  Vaccine Strain Matched V1V2 : gp70-TV1.GSKvacV1V2/293F | 12 | 0
  Vaccine Strain Matched V1V2 : gp70_C.1086C V1/V2/293F | 54 | 0

21. Secondary Outcome: Number of Participants With Occurrence of Vaccine-induced IgA Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay,run at 1:10 dilution.The readout is background-subtracted mean fluorescent intensity (MFI),with background adjustment for an antigen-specific plate level control.For each sample,response magnitude is net MFI,defined as experimental antigen MFI minus reference antigen MFI.Net MFI lt 1 is set to 1, and net MFI > 22,000 is set to 22,000.Data are excluded if blood draw date was outside the allowable window,a participant was HIV-infected,reference antigen > 5,000 MFI or baseline net MFI > 6,500.Samples from post-enrollment visits have positive responses if they meet three criteria:(1) net MFI greater than or equal to an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI),(2) net MFI values are greater than 3 times baseline net MFI, and (3) experimental antigen MFI values are greater than 3 times baseline MFI.
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 120 | 10
Participants
  Bio-1086C C1_HS | 0 | 0
  Bio-96ZM651 C1_HS | 0 | 0
  Bio-TV1 C1_HS | 0 | 0
  RV144 CoR IgA Primary gp120 Score : 00MSA 4076 gp140 | 60 | 0
  RV144 CoR IgA Primary gp120 Score : 92TH023 gp120 gDneg 293F mon | 48 | 0
  RV144 CoR IgA Primary gp120 Score : A1.con.env03 140 CF | 72 | 0
  RV144 CoR IgA Primary gp120 Score : A244 gp 120 gDneg/293F/mon | 34 | 0
  RV144 CoR IgA Primary gp120 Score : B.con.env03 140 CF | 83 | 0
  RV144 CoR IgA Primary gp120 Score : C.con.env03 140 CF_avi | 75 | 0
  RV144 CoR IgA Primary gp120 Score : Con 6 gp120/B | 68 | 0
  RV144 CoR IgA Primary gp120 Score : Con S gp140 CFI | 95 | 0
  RV144 CoR IgA Primary gp120 Score : G.con.env03 140 CF | 73 | 0
  RV144 CoR IgA Primary gp120 Score : HV 13700 AE.con.env03 140 CF | 41 | 0
  RV144 CoR IgA Primary gp120 Score : HV 14000 (DRCBL) gp140 | 65 | 0
  RV144 CoR IgA : Bio-92TH023 C1_HS | 0 | 0
  Vaccine Matched Env : 1086C_D7gp120.avi/293F | 114 | 0
  Vaccine Matched Env : 96ZM651.D11gp120.avi: number analyzed (Participants) | 120 | 9
  Vaccine Matched Env : 96ZM651.D11gp120.avi | 82 | 0
  Vaccine Matched Env : TV1c8_D11gp120.avi/293F | 90 | 0
  gp41: number analyzed (Participants) | 118 | 10
  gp41 | 0 | 0
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 118 | 10
  gp70-96ZM651.02 V1v2 | 1 | 0
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 119 | 10
  gp70-TV1.GSKvacV1V2/293F | 4 | 0
  gp70_C.1086C V1/V2/293F: number analyzed (Participants) | 109 | 10
  gp70_C.1086C V1/V2/293F | 13 | 0

22. Secondary Outcome: Level of Vaccine-induced IgG Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 and 1:100 dilutions. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI lt 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI or baseline net MFI > 6,500. Summary was calculated among positive responders only. The immune response data were also studied for their ability to predict HIV-1 infection through Month 24 (correlates of risk analysis). The comprehensive analysis results are available in Moodie et al 2022 (PubMed ID: 35758878).
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: net mean fluorescent intensity (net MFI)
Arm/Group | Vaccine
Number analyzed (Participants) | 120
net mean fluorescent intensity (net MFI)
  HVTN 505 Env Breadth Panel: VRC A_avi, dilution 1: 50: number analyzed (Participants) | 117
  HVTN 505 Env Breadth Panel: VRC A_avi, dilution 1: 50 | 20132 [8982.8 to 22000]
  HVTN 505 Env Breadth Panel: VRC A_avi, dilution 1:100: number analyzed (Participants) | 117
  HVTN 505 Env Breadth Panel: VRC A_avi, dilution 1:100 | 10290 [4369.2 to 20537.2]
  HVTN 505 Env Breadth Panel: VRC B gp140, dilution 1: 50: number analyzed (Participants) | 116
  HVTN 505 Env Breadth Panel: VRC B gp140, dilution 1: 50 | 7503.5 [4020.5 to 13312.1]
  HVTN 505 Env Breadth Panel: VRC B gp140, dilution 1:100: number analyzed (Participants) | 116
  HVTN 505 Env Breadth Panel: VRC B gp140, dilution 1:100 | 3708.5 [1640.5 to 7191.8]
  HVTN 505 Env Breadth Panel: VRC C_avi, dilution 1: 50: number analyzed (Participants) | 117
  HVTN 505 Env Breadth Panel: VRC C_avi, dilution 1: 50 | 12765 [7504.8 to 20089.5]
  HVTN 505 Env Breadth Panel: VRC C_avi, dilution 1:100: number analyzed (Participants) | 117
  HVTN 505 Env Breadth Panel: VRC C_avi, dilution 1:100 | 6247.2 [3347.5 to 11681.8]
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140, dilution 1: 50 | 17184 [9261.5 to 22000]
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140, dilution 1:100 | 8842.2 [4311.8 to 16801.8]
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon, dilution 1: 50 | 18126.8 [11247.2 to 22000]
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon, dilution 1:100 | 8697.2 [5161.8 to 16319.8]
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF, dilution 1: 50 | 22000 [19561 to 22000]
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF, dilution 1:100 | 21073.2 [10314.8 to 22000]
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi, dilution 1: 50 | 19326.2 [11303.5 to 22000]
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi, dilution 1:100 | 11210.5 [5829.5 to 17740]
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B, dilution 1: 50: number analyzed (Participants) | 114
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B, dilution 1: 50 | 15732 [9491.3 to 20903.4]
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B, dilution 1:100: number analyzed (Participants) | 114
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B, dilution 1:100 | 7617.4 [4618.9 to 11111.1]
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI, dilution 1: 50: number analyzed (Participants) | 114
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI, dilution 1: 50 | 22000 [22000 to 22000]
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI, dilution 1:100: number analyzed (Participants) | 114
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI, dilution 1:100 | 22000 [20274.6 to 22000]
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF, dilution 1: 50 | 22000 [22000 to 22000]
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF, dilution 1:100 | 22000 [14411.5 to 22000]
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF, dilution 1: 50 | 15539.5 [8042 to 22000]
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF, dilution 1:100 | 6859 [3508.2 to 14297.2]
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140, dilution 1: 50 | 10932 [6895.2 to 19457.2]
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140, dilution 1:100 | 5141.5 [2910.8 to 9346.5]
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K, dilution 1: 50: number analyzed (Participants) | 63
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K, dilution 1: 50 | 1133.8 [416.2 to 4078.9]
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K, dilution 1:100: number analyzed (Participants) | 63
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K, dilution 1:100 | 527.5 [202.1 to 1440.6]
  RV144 CoR IgG: 92TH023 gp120 gDneg 293F mon, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgG: 92TH023 gp120 gDneg 293F mon, dilution 1: 50 | 15096.5 [9387.8 to 22000]
  RV144 CoR IgG: 92TH023 gp120 gDneg 293F mon, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgG: 92TH023 gp120 gDneg 293F mon, dilution 1:100 | 7544.2 [4182.8 to 13109]
  RV144 CoR IgG: A1.con.env03 140 CF, dilution 1: 50: number analyzed (Participants) | 117
  RV144 CoR IgG: A1.con.env03 140 CF, dilution 1: 50 | 19319.5 [12159.5 to 22000]
  RV144 CoR IgG: A1.con.env03 140 CF, dilution 1:100: number analyzed (Participants) | 117
  RV144 CoR IgG: A1.con.env03 140 CF, dilution 1:100 | 12505.2 [6220.2 to 19676.2]
  RV144 CoR IgG: AE.A244 V1V2 Tags/293F, dilution 1: 50: number analyzed (Participants) | 103
  RV144 CoR IgG: AE.A244 V1V2 Tags/293F, dilution 1: 50 | 2659.8 [1054.1 to 7085.2]
  RV144 CoR IgG: AE.A244 V1V2 Tags/293F, dilution 1:100: number analyzed (Participants) | 103
  RV144 CoR IgG: AE.A244 V1V2 Tags/293F, dilution 1:100 | 1014.8 [430.4 to 2907.5]
  RV144 CoR IgG: C.1086C_V1_V2 Tags, dilution 1: 50: number analyzed (Participants) | 86
  RV144 CoR IgG: C.1086C_V1_V2 Tags, dilution 1: 50 | 1273 [525.2 to 3343.3]
  RV144 CoR IgG: C.1086C_V1_V2 Tags, dilution 1:100: number analyzed (Participants) | 86
  RV144 CoR IgG: C.1086C_V1_V2 Tags, dilution 1:100 | 566.5 [266.3 to 1335.4]
  RV144 CoR IgG: gp70-92TH023 V1V2, dilution 1: 50: number analyzed (Participants) | 112
  RV144 CoR IgG: gp70-92TH023 V1V2, dilution 1: 50 | 20359.2 [7733.3 to 22000]
  RV144 CoR IgG: gp70-92TH023 V1V2, dilution 1:100: number analyzed (Participants) | 112
  RV144 CoR IgG: gp70-92TH023 V1V2, dilution 1:100 | 7925.4 [2726.2 to 22000]
  RV144 CoR IgG: gp70_B.CaseA_V1_V2, dilution 1: 50: number analyzed (Participants) | 62
  RV144 CoR IgG: gp70_B.CaseA_V1_V2, dilution 1: 50 | 974.4 [360.8 to 3270.8]
  RV144 CoR IgG: gp70_B.CaseA_V1_V2, dilution 1:100: number analyzed (Participants) | 62
  RV144 CoR IgG: gp70_B.CaseA_V1_V2, dilution 1:100 | 452.8 [173.9 to 1350.2]
  RV144 CoR IgA: Bio-1086C C1_HS, dilution 1: 40: number analyzed (Participants) | 59
  RV144 CoR IgA: Bio-1086C C1_HS, dilution 1: 40 | 657 [324.1 to 1034.6]
  RV144 CoR IgA: Bio-92TH023 C1_HS, dilution 1: 40: number analyzed (Participants) | 96
  RV144 CoR IgA: Bio-92TH023 C1_HS, dilution 1: 40 | 3345.5 [1613.6 to 6390.6]
  RV144 CoR IgA: Bio-96ZM651 C1_HS, dilution 1: 40: number analyzed (Participants) | 92
  RV144 CoR IgA: Bio-96ZM651 C1_HS, dilution 1: 40 | 6250.6 [3556.6 to 11699.8]
  RV144 CoR IgA: Bio-TV1 C1_HS, dilution 1: 40: number analyzed (Participants) | 42
  RV144 CoR IgA: Bio-TV1 C1_HS, dilution 1: 40 | 318 [232.2 to 556.9]
  Vaccine Matched Env: 1086C_D7gp120.avi/293F, dilution 1: 50: number analyzed (Participants) | 114
  Vaccine Matched Env: 1086C_D7gp120.avi/293F, dilution 1: 50 | 22000 [22000 to 22000]
  Vaccine Matched Env: 1086C_D7gp120.avi/293F, dilution 1:100: number analyzed (Participants) | 114
  Vaccine Matched Env: 1086C_D7gp120.avi/293F, dilution 1:100 | 22000 [22000 to 22000]
  Vaccine Matched Env: 96ZM651.D11gp120.avi, dilution 1: 50: number analyzed (Participants) | 113
  Vaccine Matched Env: 96ZM651.D11gp120.avi, dilution 1: 50 | 22000 [22000 to 22000]
  Vaccine Matched Env: 96ZM651.D11gp120.avi, dilution 1:100: number analyzed (Participants) | 113
  Vaccine Matched Env: 96ZM651.D11gp120.avi, dilution 1:100 | 19310.5 [12406.2 to 22000]
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F, dilution 1: 50: number analyzed (Participants) | 114
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F, dilution 1: 50 | 22000 [22000 to 22000]
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F, dilution 1:100: number analyzed (Participants) | 114
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F, dilution 1:100 | 22000 [22000 to 22000]
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2, dilution 1: 50: number analyzed (Participants) | 61
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2, dilution 1: 50 | 1319.8 [620 to 4714.8]
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2, dilution 1:100: number analyzed (Participants) | 61
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2, dilution 1:100 | 538.5 [283.8 to 1248.8]
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F, dilution 1: 50: number analyzed (Participants) | 73
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F, dilution 1: 50 | 1452.8 [530.2 to 5018.2]
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F, dilution 1:100: number analyzed (Participants) | 73
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F, dilution 1:100 | 640.2 [259.5 to 1809.5]
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F, dilution 1: 50: number analyzed (Participants) | 103
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F, dilution 1: 50 | 4573.2 [1793.4 to 14216.1]
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F, dilution 1:100: number analyzed (Participants) | 103
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F, dilution 1:100 | 2029.2 [688.2 to 6273.9]
  gp41, dilution 1: 50: number analyzed (Participants) | 1
  gp41, dilution 1: 50 | 2125 [2125 to 2125]
  gp41, dilution 1:100: number analyzed (Participants) | 1
  gp41, dilution 1:100 | 780.8 [780.8 to 780.8]

23. Secondary Outcome: Level of Vaccine-induced IgG3 Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgG3 responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:40 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI lt 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI or baseline net MFI > 6,500. Summary was calculated among positive responders only. The immune response data were also studied for their ability to predict HIV-1 infection through Month 24 (correlates of risk analysis). The comprehensive analysis results are available in Moodie et al 2022 (PubMed ID: 35758878).
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: net mean fluorescent intensity (net MFI)
Arm/Group | Vaccine
Number analyzed (Participants) | 120
net mean fluorescent intensity (net MFI)
  HVTN 505 Env Breadth Panel: A1.con.env03 140 CF: number analyzed (Participants) | 74
  HVTN 505 Env Breadth Panel: A1.con.env03 140 CF | 277.1 [171.1 to 702.7]
  HVTN 505 Env Breadth Panel: B.con.env03 140 CF: number analyzed (Participants) | 106
  HVTN 505 Env Breadth Panel: B.con.env03 140 CF | 369.5 [217.2 to 974.2]
  HVTN 505 Env Breadth Panel: C.con.env03 140 CF_avi: number analyzed (Participants) | 87
  HVTN 505 Env Breadth Panel: C.con.env03 140 CF_avi | 302.2 [154.2 to 601.5]
  HVTN 505 Env Breadth Panel: Con 6 gp120/B: number analyzed (Participants) | 99
  HVTN 505 Env Breadth Panel: Con 6 gp120/B | 318.5 [181.5 to 775.5]
  HVTN 505 Env Breadth Panel: Con S gp140 CFI: number analyzed (Participants) | 115
  HVTN 505 Env Breadth Panel: Con S gp140 CFI | 843 [471.9 to 2435]
  HVTN 505 Env Breadth Panel: VRC A_avi: number analyzed (Participants) | 72
  HVTN 505 Env Breadth Panel: VRC A_avi | 337.8 [160.2 to 844.6]
  HVTN 505 Env Breadth Panel: VRC B gp140: number analyzed (Participants) | 42
  HVTN 505 Env Breadth Panel: VRC B gp140 | 208.2 [140.9 to 432.4]
  HVTN 505 Env Breadth Panel: VRC C_avi: number analyzed (Participants) | 68
  HVTN 505 Env Breadth Panel: VRC C_avi | 262.9 [135.2 to 540.8]
  RV144 CoR IgG3: C.1086C_V1_V2 Tags: number analyzed (Participants) | 32
  RV144 CoR IgG3: C.1086C_V1_V2 Tags | 277.5 [131.2 to 601.6]
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K: number analyzed (Participants) | 9
  RV144 CoR IgG3: gp70_B.CaseA2 V1/V2/169K | 963.5 [213.8 to 3295.5]
  RV144 CoR IgG3: gp70_B.CaseA_V1_V2: number analyzed (Participants) | 8
  RV144 CoR IgG3: gp70_B.CaseA_V1_V2 | 1598.9 [316.9 to 3041.8]
  V1V2 Subtype AW: AE.A244 V1V2 Tags/293F: number analyzed (Participants) | 49
  V1V2 Subtype AW: AE.A244 V1V2 Tags/293F | 350.8 [237 to 868.8]
  Vaccine Matched Env: 1086C_D7gp120.avi/293F | 4534.8 [2132.6 to 11252.6]
  Vaccine Matched Env: 96ZM651.D11gp120.avi: number analyzed (Participants) | 110
  Vaccine Matched Env: 96ZM651.D11gp120.avi | 700.5 [333.9 to 1815.9]
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 118
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F | 2059.5 [896.6 to 5165.4]
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2: number analyzed (Participants) | 10
  Vaccine Strain Matched V1V2: gp70-96ZM651.02 V1v2 | 1398.2 [370.2 to 3796.9]
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 12
  Vaccine Strain Matched V1V2: gp70-TV1.GSKvacV1V2/293F | 511.4 [222.6 to 1469.4]
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F: number analyzed (Participants) | 54
  Vaccine Strain Matched V1V2: gp70_C.1086C V1/V2/293F | 572.6 [379.7 to 1367.2]

24. Secondary Outcome: Level of Vaccine-induced IgA Binding Antibodies to HIV Proteins at Month 6.5
Description: Serum IgA responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:10 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Net MFI lt 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI or baseline net MFI > 6,500. Summary was calculated among positive responders only. The immune response data were also studied for their ability to predict HIV-1 infection through Month 24 (correlates of risk analysis). The comprehensive analysis results are available in Moodie et al 2022 (PubMed ID: 35758878).
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: net mean fluorescent intensity (net MFI)
Arm/Group | Vaccine
Number analyzed (Participants) | 120
net mean fluorescent intensity (net MFI)
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140: number analyzed (Participants) | 60
  RV144 CoR IgA Primary gp120 Score: 00MSA 4076 gp140 | 1521.5 [657.8 to 3967.9]
  RV144 CoR IgA Primary gp120 Score: 92TH023 gp120 gDneg 293F mon: number analyzed (Participants) | 48
  RV144 CoR IgA Primary gp120 Score: 92TH023 gp120 gDneg 293F mon | 1024.8 [666.6 to 1453.9]
  RV144 CoR IgA Primary gp120 Score: A1.con.env03 140 CF: number analyzed (Participants) | 72
  RV144 CoR IgA Primary gp120 Score: A1.con.env03 140 CF | 2511.9 [949.1 to 5347]
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon: number analyzed (Participants) | 34
  RV144 CoR IgA Primary gp120 Score: A244 gp 120 gDneg/293F/mon | 801.2 [506.3 to 1325.8]
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF: number analyzed (Participants) | 83
  RV144 CoR IgA Primary gp120 Score: B.con.env03 140 CF | 3140.2 [1685 to 6907.4]
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi: number analyzed (Participants) | 75
  RV144 CoR IgA Primary gp120 Score: C.con.env03 140 CF_avi | 2149.8 [1102.6 to 4907]
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B: number analyzed (Participants) | 68
  RV144 CoR IgA Primary gp120 Score: Con 6 gp120/B | 2877.9 [1620.6 to 5074.7]
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI: number analyzed (Participants) | 95
  RV144 CoR IgA Primary gp120 Score: Con S gp140 CFI | 5239.2 [2974.8 to 11492.1]
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF: number analyzed (Participants) | 73
  RV144 CoR IgA Primary gp120 Score: G.con.env03 140 CF | 2845 [1261 to 6844.8]
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF: number analyzed (Participants) | 41
  RV144 CoR IgA Primary gp120 Score: HV 13700 AE.con.env03 140 CF | 791 [483.8 to 1970.2]
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140: number analyzed (Participants) | 65
  RV144 CoR IgA Primary gp120 Score: HV 14000 (DRCBL) gp140 | 1291.5 [588.2 to 3242]
  Vaccine Matched Env: 1086C_D7gp120.avi/293F: number analyzed (Participants) | 114
  Vaccine Matched Env: 1086C_D7gp120.avi/293F | 22000 [21620.4 to 22000]
  Vaccine Matched Env: 96ZM651.D11gp120.avi: number analyzed (Participants) | 82
  Vaccine Matched Env: 96ZM651.D11gp120.avi | 6673.8 [4418.9 to 10935.2]
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F: number analyzed (Participants) | 90
  Vaccine Matched Env: TV1c8_D11gp120.avi/293F | 6205 [3399 to 9946.1]
  gp70-96ZM651.02 V1v2: number analyzed (Participants) | 1
  gp70-96ZM651.02 V1v2 | 22000 [22000 to 22000]
  gp70-TV1.GSKvacV1V2/293F: number analyzed (Participants) | 4
  gp70-TV1.GSKvacV1V2/293F | 1059.5 [731.9 to 3515.9]
  gp70_C.1086C V1/V2/293F: number analyzed (Participants) | 13
  gp70_C.1086C V1/V2/293F | 5786.5 [5169 to 8446]

25. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through 24 Months Among Female Participants
Description: Vaccine efficacy was calculated as 1 minus the hazard ratio for HIV-1 infection, which was estimated using a Cox proportional-hazards (Cox PH) model and tested using a log-rank test.
Time Frame: Measured through 24 months after first vaccination
Population: Females in MITT cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1887 | 1886
events per 100 person-years | 0.043 | 0.042
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.82, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.80 to 1.33] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through 24 Months Among Male Participants
Description: as for outcome 25
Time Frame: Measured through 24 months after first vaccination
Population: Males in MITT cohort
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 808 | 803
events per 100 person-years | 0.013 | 0.013
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.98, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.50 to 1.98] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through 24 Months Among Female Participants Aged 25 or Younger
Description: as for outcome 25
Time Frame: Measured through 24 months after first vaccination
Population: Females in MITT cohort aged 25 or younger
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1264 | 1267
events per 100 person-years | 0.047 | 0.044
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.60, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.80 to 1.47] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through 24 Months Among Female Participants Older Than 25
Description: as for outcome 25
Time Frame: Measured through 24 months after first vaccination
Population: Females in MITT cohort older than 25
Measure: Number; unit: events per 100 person-years
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 623 | 619
events per 100 person-years | 0.035 | 0.039
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.71, Log Rank; The hazard ratio was tested using a sex-stratified log rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.58 to 1.46] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Incidence Rate of HIV-1 Infection Diagnosed After Enrollment Through Month 24 by Genotypic Characteristics of Viral Sequences From HIV-1 Infected Participants at HIV-1 Diagnosis, Such As Signature Site Mutations
Description: Analysis will only be performed if significant positive evidence of vaccine efficacy from enrollment through 24 months is seen. However, monitoring boundaries for non-efficacy have been met per the 23 January 2020 DSMB finding.
Time Frame: Measured through 24 months after first vaccination
Population: Analysis will only be performed if significant positive evidence of vaccine efficacy from enrollment through 24 months is seen. However, monitoring boundaries for non-efficacy have been met per the 23 January 2020 DSMB finding.
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Number of Participants With Viral Sequences at HIV-1 Diagnosis
Description: Number of participants in the female mITT cohort with viral sequences were reported. Viral sequencing was conducted on the earliest available plasma specimens with positive HIV-1 RNA PCR tests from study participants who are diagnosed with HIV-1 infection.
Time Frame: Measured through 24 months after first vaccination
Population: The female mITT cohort was the group of participants used in sieve analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 122 | 117
Participants | 119 | 115

ADVERSE EVENTS:
Time Frame: Serious adverse events, adverse events of special interest, adverse events of STIs, new chronic medical conditions, and adverse events leading to early participant withdrawal or early discontinuation of study product(s) administration were collected through 12 months after the last vaccination received. All other adverse events were collected through 30 days after each vaccination.
Description: Adverse events of special interest (AESI) were described in Appendix J of the protocol. AESI for this protocol include but are not limited to potential immune-mediated diseases.
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 8/2704 | 10/2700
Serious Adverse Events (participants affected / at risk) | 103/2704 | 95/2700
Other Adverse Events (participants affected / at risk) | 1707/2704 | 1704/2700
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=2704) | Placebo (N=2700)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Any Event in SOC (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Any Event in SOC (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 3 (3) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Any Event in SOC (General disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Electrocution (General disorders) | 1 (1) | 0 (0)
Mass (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Any Event in SOC (Hepatobiliary disorders) | 4 (6) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (2) | 0 (0)
Any Event in SOC (Infections and infestations) | 15 (16) | 17 (20)
Abscess limb (Infections and infestations) | 0 (0) | 2 (2)
Acute hepatitis B (Infections and infestations) | 0 (0) | 2 (2)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Genital abscess (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 42 (44) | 38 (40)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Any Event in SOC (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 5 (5) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 12 (12)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (4)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 11 (11) | 12 (12)
Acute psychosis (Psychiatric disorders) | 0 (0) | 2 (2)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 3 (3)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 2 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 4 (4) | 1 (1)
Any Event in SOC (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Any Event in SOC (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=2704) | Placebo (N=2700)
Any Event in SOC (Blood and lymphatic system disorders) | 11 (12) | 11 (12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 9 (9) | 5 (5)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Any Event in SOC (Cardiac disorders) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 10 (10) | 3 (3)
Cerumen impaction (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Any Event in SOC (Endocrine disorders) | 0 (0) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Any Event in SOC (Eye disorders) | 17 (18) | 16 (16)
Atopic keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 5 (5) | 9 (9)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 4 (4) | 0 (0)
Eye pruritus (Eye disorders) | 2 (2) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Periorbital pain (Eye disorders) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 1 (1) | 0 (0)
Photokeratitis (Eye disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 151 (165) | 162 (178)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 22 (22) | 18 (18)
Abdominal pain lower (Gastrointestinal disorders) | 10 (10) | 15 (15)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 5 (5)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (8) | 3 (3)
Dental caries (Gastrointestinal disorders) | 7 (7) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 29 (29) | 41 (44)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 10 (10)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 15 (15) | 11 (12)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 5 (6)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 9 (9)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 2 (3)
Mouth cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 11 (11)
Peptic ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 17 (17) | 10 (10)
Vomiting (Gastrointestinal disorders) | 8 (8) | 11 (11)
Any Event in SOC (General disorders) | 206 (233) | 198 (218)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 2 (4) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 6 (6) | 9 (9)
Hangover (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 166 (181) | 171 (188)
Injection site bruising (General disorders) | 2 (2) | 1 (1)
Injection site dermatitis (General disorders) | 0 (0) | 1 (1)
Injection site discolouration (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3)
Injection site pruritus (General disorders) | 21 (23) | 2 (2)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Injection site ulcer (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1)
Mass (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Any Event in SOC (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Any Event in SOC (Immune system disorders) | 4 (4) | 3 (3)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Any Event in SOC (Infections and infestations) | 1243 (2247) | 1295 (2290)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 8 (9) | 11 (11)
Acarodermatitis (Infections and infestations) | 36 (37) | 34 (37)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Bacterial urethritis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 5 (5) | 7 (7)
Bartholin's abscess (Infections and infestations) | 3 (3) | 2 (2)
Body tinea (Infections and infestations) | 17 (17) | 23 (24)
Bronchitis (Infections and infestations) | 4 (4) | 6 (6)
Cellulitis (Infections and infestations) | 2 (2) | 6 (6)
Cestode infection (Infections and infestations) | 0 (0) | 1 (1)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 3 (3) | 2 (2)
Chronic hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 8 (8) | 7 (7)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 3 (3)
Dysentery (Infections and infestations) | 0 (0) | 3 (3)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Ecthyma (Infections and infestations) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 20 (20) | 9 (9)
Fungal skin infection (Infections and infestations) | 11 (12) | 6 (6)
Furuncle (Infections and infestations) | 1 (1) | 4 (5)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 46 (50) | 53 (57)
Gastroenteritis viral (Infections and infestations) | 10 (10) | 9 (9)
Genital abscess (Infections and infestations) | 2 (2) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 3 (4)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Genital ulcer syndrome (Infections and infestations) | 8 (8) | 20 (23)
Genitourinary chlamydia infection (Infections and infestations) | 661 (908) | 689 (917)
Genitourinary tract gonococcal infection (Infections and infestations) | 286 (332) | 272 (319)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 2 (2) | 4 (5)
Gonococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 2 (2)
Impetigo (Infections and infestations) | 9 (9) | 3 (3)
Implant site abscess (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 7 (7)
Injection site cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Joint abscess (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1)
Latent syphilis (Infections and infestations) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 27 (27) | 18 (20)
Lymphogranuloma venereum (Infections and infestations) | 0 (0) | 2 (2)
Male genital tract tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Nasal abscess (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 10 (10)
Omphalitis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 11 (11) | 2 (2)
Oral pustule (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 4 (4)
Otitis externa (Infections and infestations) | 3 (3) | 4 (4)
Otitis media (Infections and infestations) | 4 (4) | 2 (2)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 12 (12) | 6 (7)
Pharyngitis (Infections and infestations) | 10 (10) | 8 (8)
Pharyngotonsillitis (Infections and infestations) | 1 (2) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 27 (32) | 13 (18)
Proctitis gonococcal (Infections and infestations) | 10 (10) | 12 (13)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 11 (12)
Pustule (Infections and infestations) | 3 (3) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 5 (5) | 5 (6)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 10 (10) | 10 (11)
Schistosomiasis (Infections and infestations) | 1 (1) | 1 (1)
Secondary syphilis (Infections and infestations) | 1 (1) | 1 (2)
Sexually transmitted disease (Infections and infestations) | 6 (6) | 2 (2)
Sinusitis (Infections and infestations) | 7 (8) | 3 (3)
Skin bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 24 (26) | 26 (27)
Syphilis (Infections and infestations) | 41 (46) | 34 (38)
Syphilis genital (Infections and infestations) | 1 (1) | 2 (2)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 3 (3) | 1 (1)
Tinea faciei (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 2 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Tinea versicolour (Infections and infestations) | 12 (13) | 12 (12)
Tonsillitis (Infections and infestations) | 31 (33) | 34 (35)
Tonsillitis bacterial (Infections and infestations) | 2 (2) | 3 (3)
Tooth abscess (Infections and infestations) | 3 (3) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 131 (142) | 119 (127)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urethritis (Infections and infestations) | 25 (28) | 31 (35)
Urinary tract infection (Infections and infestations) | 47 (50) | 50 (53)
Urinary tract infection bacterial (Infections and infestations) | 4 (4) | 8 (8)
Urogenital trichomoniasis (Infections and infestations) | 6 (6) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 3 (3)
Vaginitis chlamydial (Infections and infestations) | 7 (7) | 2 (2)
Varicella (Infections and infestations) | 0 (0) | 2 (2)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibulitis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 3 (3) | 5 (5)
Viral pharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Viral sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Viral tonsillitis (Infections and infestations) | 1 (1) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 14 (14) | 22 (23)
Vulval abscess (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 33 (37) | 38 (39)
Vulvovaginitis (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginitis chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginitis gonococcal (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 150 (179) | 165 (210)
Wound infection (Infections and infestations) | 1 (1) | 2 (2)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 118 (124) | 80 (84)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
First degree chemical burn of skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body in ear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Genital contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Herbal toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 11 (11) | 5 (5)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 13 (13) | 6 (6)
Lip injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
Neck injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 13 (13) | 10 (10)
Soft tissue injury (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Stab wound (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 8 (8) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 92 (108) | 95 (111)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 47 (59) | 53 (63)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 3 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 38 (42) | 38 (44)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 24 (25) | 20 (20)
Abnormal loss of weight (Metabolism and nutrition disorders) | 11 (11) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 90 (95) | 98 (106)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 20 (20)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (26) | 29 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 5 (5)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 11 (11)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (14) | 13 (13)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 8 (8)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Any Event in SOC (Nervous system disorders) | 165 (178) | 151 (166)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 24 (25) | 22 (22)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 117 (121) | 107 (114)
Migraine (Nervous system disorders) | 1 (1) | 3 (3)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Sensory loss (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 5 (5)
Tension headache (Nervous system disorders) | 15 (16) | 10 (10)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Product Issues) | 0 (0) | 1 (1)
Device expulsion (Product Issues) | 0 (0) | 1 (1)
Any Event in SOC (Psychiatric disorders) | 17 (19) | 20 (22)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (5)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1)
Loss of libido (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1) | 1 (1)
Substance-induced mood disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 20 (21) | 23 (23)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 8 (8)
Haematuria (Renal and urinary disorders) | 1 (1) | 5 (5)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 12 (12) | 6 (6)
Urethral discharge (Renal and urinary disorders) | 2 (2) | 2 (2)
Urethral syndrome (Renal and urinary disorders) | 2 (2) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 167 (190) | 176 (193)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 5 (5) | 7 (7)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile blister (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 134 (154) | 132 (142)
Vulval ulceration (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3) | 8 (8)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 53 (55) | 40 (42)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 13 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (15)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 136 (147) | 134 (146)
Acne (Skin and subcutaneous tissue disorders) | 13 (13) | 7 (7)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 12 (12) | 12 (12)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (22) | 22 (23)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 15 (15) | 24 (24)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 17 (17) | 13 (16)
Rash pruritic (Skin and subcutaneous tissue disorders) | 15 (15) | 11 (12)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Any Event in SOC (Social circumstances) | 1 (1) | 2 (2)
Physical assault (Social circumstances) | 0 (0) | 1 (1)
Victim of sexual abuse (Social circumstances) | 1 (1) | 1 (1)
Any Event in SOC (Vascular disorders) | 24 (29) | 21 (23)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 21 (26) | 17 (19)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT02968849/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT02968849/SAP_001.pdf